CLINICAL TRIAL: NCT05451485
Title: Vector Flow Imaging in Healthy Vessels
Brief Title: VFI in Healthy Vessels
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NL80478.091.22
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Carotid Artery Stenosis; Superficial Femoral Artery Stenosis
Keywords: Vector Flow Imaging; Ultrasound Particle Image Velocimetry; Blood Speckle Tracking; 4D flow MR
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young volunteers: Volunteers with age between 20-30 years
  Interventions: Diagnostic Test: Blood speckle tracking; Diagnostic Test: Ultrasound particle Imaging Velocimetry; Diagnostic Test: 4D flow MRI; Diagnostic Test: Conventional duplex
- Old volunteers: Volunteers with age between 65-75 years
  Interventions: Diagnostic Test: Blood speckle tracking; Diagnostic Test: Ultrasound particle Imaging Velocimetry; Diagnostic Test: 4D flow MRI; Diagnostic Test: Conventional duplex

INTERVENTIONS:
Diagnostic Test: Blood speckle tracking — Blood speckle tracking measurements will be acquired of the carotid artery and superficial femoral artery
Diagnostic Test: Ultrasound particle Imaging Velocimetry — Ultrasound particle imaging velocimetry will be acquired of the carotid artery and superficial femoral artery
Diagnostic Test: 4D flow MRI — 4D flow MRI will be acquired of the carotid artery and superficial femoral artery
Diagnostic Test: Conventional duplex — Conventional duplex measurements will be acquired of the carotid artery and superficial femoral artery

SUMMARY:
There is a wealth of evidence implicating the important role of blood flow throughout all stages of the process of atherogenesis. Two locations along the vascular tree at which atherosclerotic plaques are typically found are the carotid artery (CA) and the superficial femoral artery (SFA). Nowadays, ultrasound is the technique of choice for assessing the vascular condition in the CA and SFA. However, clinically used ultrasound techniques show a large variability in estimating the blood flow velocity, due to multiple limitations. With the advent of ultrafast ultrasound imaging, (almost) all elements of the transducer can be activated simultaneously. These so-called plane wave acquisition acquires thousands of images per second and makes continuous tracking of blood flow velocities in all directions in the field of view possible. This high-frame-rate acquisition opened up new possibilities for blood flow imaging at the CA and SFA, such as blood Speckle Tracking (bST) and ultrasound Particle Image Velocimetry (echoPIV). Both these vector flow imaging (VFI) techniques enable the quantification of 2D blood flow velocity profiles, where bST uses no contrast agents compared to echoPIV. Beside these novel ultrasound based techniques, 4D Phase Contrast Magnetic Resonance Imaging (4D flow MRI) enables a non-invasive quantification of the 4D blood flow velocity profiles (3D + time) and can be used as reference standard for blood flow assessments in-vivo. We therefore aim to evaluate the performance of both VFI techniques in comparison to 4D flow MRI measurements in the CA and SFA of healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female, without cardiovascular and pulmonary medical history and without the use of medication for cardiovascular risk factors
* Age between 20-30 year or 65-75 years old
* Willingness to undergo a 4D flow MRI scan and US examinations
* Informed consent form understood and signed, and agrees to the hospital visit

Exclusion Criteria:

* Hypersensitivity to the active substance(s) or any of the excipients in Sonovue
* Pregnancy
* MRI exclusion criteria (such as presence of pacemaker, cerebral vascular clips, claustrophobia)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Both young (n=10) and old (n=10) groups will exist of five female and five male subjects.
Study Population: The study population will include twenty healthy subjects divided in two different age groups.
  All volunteers will be recruited within Rijnstate hospital and Radboudumc.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-11-05 (Actual); Primary Completion 2023-03-18 (Actual); Study Completion 2023-03-18 (Actual)

PRIMARY OUTCOMES:
Validation VFI with MRI (echoPIV) | 1 day (no follow-up)
  Two-dimensional vector velocity fields derived from VFI (echoPIV) and 4D flow MRI will be used to calculate the spatiotemporal blood flow velocity profiles in artery
Validation VFI with MRI (bST) | 1 day (no follow-up)
  Two-dimensional vector velocity fields derived from VFI (bST) and 4D flow MRI will be used to calculate the spatiotemporal blood flow velocity profiles in artery

SECONDARY OUTCOMES:
Correlation VFI techniques (bST vs echoPIV) | 1 day (no follow-up)
  Two-dimensional vector velocity fields derived from echoPIV and bST will be used to calculate the spatiotemporal blood flow velocity profiles in the artery
Flow derived parameters (WSS) | 1 day (no follow-up)
  Two-dimensional vector velocity fields derived from VFI and 4D flow MRI will be used to calculate the flow derived parameters in the artery. Multiple flow derived parameters will be derived from the vector velocity data. One of the flow derived parameters is wall shear stress (WSS), which defines the amount of friction of the blood on the vessel wall.
Flow derived parameters (vorticity) | 1 day (no follow-up)
  Two-dimensional vector velocity fields derived from VFI and 4D flow MRI will be used to calculate the flow derived parameters in the artery. Multiple flow derived parameters will be derived from the vector velocity data. One of the flow derived parameters is the vorticity, or the curl of the velocity. The vorticity represents the rotation of particles inside the flow field. This measure can potentially be used to define regions with disturbed blood flow, as a high value (in rad/s) indicates the occurence of a recirculation.
Flow derived parameters (vector complexity) | 1 day (no follow-up)
  Two-dimensional vector velocity fields derived from VFI and 4D flow MRI will be used to calculate the flow derived parameters in the artery. Multiple flow derived parameters will be derived from the vector velocity data. One of the flow derived parameters is vector complexity, which is a measure of multi-directional flow, ranging from 0 till 1. a value of 1 means complex flow with all velocity vectors pointing in all directions, whereas a value of 0 means laminar flow with all velocity vectors pointing in the same direction. This measure can potentially be used to indicate regions with disturbed blood flow.
Old versus young (blood flow velocity profiles) | 1 day (no follow-up)
  Two-dimensional vector velocity fields derived from VFI and 4D flow MRI will be used to calculate the spatiotemporal blood flow velocity profiles between young and old volunteers.
Old versus young (WSS) | 1 day (no follow-up)
  Two-dimensional vector velocity fields derived from VFI and 4D flow MRI will be used to calculate different flow derived parameters between young and old volunteers. One of the parameters is WSS.
Old versus young (vector complexity) | 1 day (no follow-up)
  Two-dimensional vector velocity fields derived from VFI and 4D flow MRI will be used to calculate different flow derived parameters between young and old volunteers. One of the parameters is vector complexity.
Old versus young (vorticity) | 1 day (no follow-up)
  Two-dimensional vector velocity fields derived from VFI and 4D flow MRI will be used to calculate different flow derived parameters between young and old volunteers. One of the parameters is vorticity.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Reijnen, MD, Prof, Principal Investigator — Rijnstate Hospital
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands

REFERENCES:
- [Derived] Ruisch J, de Bakker JMK, van Helvert M, Schoonbrood MJP, Groot Jebbink E, Holewijn S, Reijnen MMPJ, de Korte CL, Saris AECM. Ultrasound-based Velocity Vector Imaging in the Carotid Bifurcation: Repeatability and an In Vivo Comparison With 4-D Flow MRI. Ultrasound Med Biol. 2025 Jun;51(6):969-976. doi: 10.1016/j.ultrasmedbio.2025.02.008. Epub 2025 Mar 6. PMID 40055083